CLINICAL TRIAL: NCT00406250
Title: Intravitreal Bevacizumab for Choroidal Neovascularization Secondary to Angioid Streaks: 24 Months Follow-up
Brief Title: Intravitreal Bevacizumab in Agioid Streaks
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Chiosi Flavia, Chiosi Flavia, University of Campania Luigi Vanvitelli
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 81612
Record Dates: First submitted 2006-11-30; First posted 2006-12-04 (Estimated); Last update posted 2016-02-08 (Estimated); Status verified 2016-02

CONDITIONS: Angioid Streaks; Choroidal Neovascularization
MeSH Terms: conditions — Angioid Streaks; Choroidal Neovascularization | interventions — Intravitreal Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bevacizumab (Experimental)
  Interventions: Drug: intravitreal injection

INTERVENTIONS:
Drug: intravitreal injection — 1.25 mg in 0.05 cc of bevacizumab
  Other Names: intravitreal bevacizumab
Drug: intravitreal injection — 1.25 mg of bevacizumab intravitreally injected in a steril field
  Other Names: intravitreal bevacizumab

SUMMARY:
The purpose of this study is to investigate the safety and efficacy of intravitreal bevacizumab in patients with choroidal neovascularization associated with angioid streaks.

DETAILED DESCRIPTION:
To investigate the safety and efficacy of intravitreal bevacizumab in a patient with choroidal neovascularization associated with angioid streaks. One of the most serious ocular complication of angioid streaks is the occurrence of choroidal neovascularization (CNV) and because of the implication of the macula, this complication usually leads to central vision loss.

During the past, laser photocoagulation, first, and photodynamic therapy (PDT), more recently, have been used as treatment for this kind of CNV. The outcome of these therapies was often variable and sometimes disappointing for the stabilization of visual acuity and lesion size in CNV secondary to AS.

Five patients (six eyes) with CNV secondary to AS participated in this retrospective interventional case series. All patients were scheduled for three monthly IVB injections (1.25 mg). Two eyes had been previously treated with photodynamic therapy (PDT), and four received IVB as first choice treatment. IVB was repeated in case of recurrence after the three monthly IVB schedule. Ophthalmic evaluations included: best corrected visual acuity (BCVA) determination (ETDRS), optical coherence tomography (OCT), fluorescein and indocyanine green angiographies. Main outcome measures were BCVA improvement, reduction of leakage from CNV and diminution of central retinal thickness (CRT). Patients were followed-up for 30 months. Patients were 3 males and 2 females aged 44 to 67 years (mean 51.6 +/- 9.07 SD), who received a mean number of 4.33 IB treatments (+/-1.5; min: 3, max: 7). The mean retreatment interval was 3 months (+/-1.36; min: 2, max: 6).

Four eyes (66.6%) showed a BCVA improvement (mean 3.4 lines) from baseline and two eyes (33.3%) did not show any change in visual acuity from baseline to last follow-up. Mean BCVA rose significantly from 22.5+/-14.4 letters at baseline to 35.8+/-21.5 letters at 30 months (p=0.025). Angiographic examinations showed reduction or cessation of the CNV leakage in all patients. OCT findings demonstrated slight CRT diminution (mean 41.6 µm). No intraocular pressure changes were observed after the IVB injection, which did not cause any systemic complication. No injection related back pain or IVB-induced ocular complication was reported.

ELIGIBILITY:
Inclusion Criteria:

* presence of an active CNV
* visual loss
* increased retinal thickness

Exclusion Criteria:

* no actively leaking CNV by FAG
* normal retinal thickness
* satisfactory visual acuity

Ages: 44 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2006-11; Primary Completion 2008-12 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
BCVA improvement | 6 months

SECONDARY OUTCOMES:
reduction or cessation leakage | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Michele Rinaldi, MD, Principal Investigator — University of Campania Luigi Vanvitelli
Locations (1):
- Dipartimento di Oftalmologia, SUN, Napoli, Napoli, Italy